CLINICAL TRIAL: NCT02143635
Title: A Phase I, Open Label, Multicenter, Dose-escalation Study of HDM201 in Adult Patients With Advanced Solid and Hematological Tumors Characterized by Wild-type TP53
Brief Title: Study to Determine and Evaluate a Safe and Tolerated Dose of HDM201 in Patients With Selected Advanced Tumors That Are TP53wt
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHDM201X2101
Record Dates: First submitted 2014-05-19; First posted 2014-05-21 (Estimated); Last update posted 2021-05-21 (Actual); Status verified 2021-05

CONDITIONS: Advanced Solid and Hematological TP53wt Tumors
Keywords: HDM201,TP53wt, p53, MDM2, HDM2, advanced tumors, BLRM (Bayesian logistic regression model)
MeSH Terms: interventions — siremadlin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Arm A (Experimental)
  Interventions: Drug: HDM201; Drug: ancillary treatment
- Arm B (Experimental)
  Interventions: Drug: HDM201
- Arm C (Experimental)
  Interventions: Drug: HDM201
- Arm D (Experimental)
  Interventions: Drug: HDM201

INTERVENTIONS:
Drug: HDM201
Drug: ancillary treatment
  Arms: Arm A

SUMMARY:
To determine and evaluate a safe and tolerated dose of HDM201 in adult patients with selected advanced tumors characterized by wild-type TP53.

ELIGIBILITY:
Inclusion Criteria:

* Patient with a TP53wt locally advanced or metastatic solid malignancy and with measurable or non-measurable (but evaluable) disease as determined by RECIST 1.1 criteria.
* Patients with the TP53wt hematological tumors (AML, ALL, HR-MDS) who have failed prior therapies or who are considered inappropriate candidates for standard induction therapy.

Other protocol-defined inclusion criteria may apply

Exclusion Criteria:

* Prior treatment with compounds with the same mode of action
* Subjects with significant or uncontrolled cardiovascular disease
* History of thromboembolic or cerebrovascular events within the last 6 months, including transient ischemic attack, cerebrovascular accident, deep vein thrombosis, or pulmonary embolism
* Previous and concomitant therapy that precludes enrollment, as defined in the protocol
* Known Human Immunodeficiency Virus (HIV) infection and/or active Hepatitis B or Hepatitis C infection
* Patients who have undergone major surgery within the 2 weeks prior to starting study treatment or who have not fully recovered from previous surgery
* Women of child-bearing potential, unless they are using highly effective methods of contraception during dosing and for 2 weeks after study drug discontinuation
* Pregnant or nursing women

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Actual)
Dates: Start 2014-07-07 (Actual); Primary Completion 2017-06-20 (Actual); Study Completion 2020-06-09 (Actual)

PRIMARY OUTCOMES:
Incidence of dose limiting toxicities (DLTs) | up to 28 days
  DLTs in the first cycle of treatment.

SECONDARY OUTCOMES:
Number of patients with adverse events (AEs) | For the duration of treatment, an average of 16 weeks
  Number of patients with AEs as a measure of Safety and tolerability of HDM201 single agent.
Pharmacokinetics (PK) parameters of HDM201 | Up to 42 days
Changes from baseline of Pharmacodynamics markers | Baseline, up to 28 days
Tumor response | Every 8 weeks (for solid tumors), every cycle (for hematological tumors) until end of treatment
  end of treatment = 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (14):
- United States (2):
  - Dana Farber Cancer Institute SC-6, Boston, Massachusetts
  - Memorial Sloan Kettering Onc. Dep, New York, New York
- France (2):
  - Novartis Investigative Site, Lyon
  - Novartis Investigative Site, Paris
- Germany (3):
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Würzburg
- Japan (2):
  - Novartis Investigative Site, Kobe, Hyōgo
  - Novartis Investigative Site, Chuo Ku, Tokyo
- Netherlands (2):
  - Novartis Investigative Site, Amsterdam
  - Novartis Investigative Site, Utrecht
- Novartis Investigative Site, Singapore, Singapore
- Novartis Investigative Site, Barcelona, Catalonia, Spain
- Novartis Investigative Site, Taipei, Taiwan ROC, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Study Results — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=17828